CLINICAL TRIAL: NCT05572359
Title: Effect of Cryo- and Compression Therapy After Total Knee and Unicompartmental Arthroplasty, A Randomised Controlled Trial
Brief Title: Cryo and Compression Therapy After TKA and UKA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Martini Hospital Groningen (Other)
Collaborators: U-sport (Unknown); Dutch Arthroplasty Register (LROI) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Record Dates: First submitted 2022-10-03; First posted 2022-10-07 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Osteo Arthritis Knee
Keywords: total knee arthroplasty; unicompartmental knee arthroplasty

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated to receive either cryo- and compression therapy during the first six weeks after surgery or standard care.
Who Masked: Outcomes Assessor
Masking Description: During the baseline visit the preoperative questionnaires will be obtained from the patient and the physical examination tests will be performed. Only after this is finished, at the end of this visit, the randomisation will be performed by opening a sealed envelope.
  All patients will be invited for a study control visit after 6 weeks. During the appointment a blinded assessor (not one of the researchers involved in the baseline measurements) will first perform the physical examination tests, after which a check of the completeness of the questionnaires will be done. Finally, the log will be checked. Patients are instructed not to talk about the intervention they received until the log was checked. In this way the preceding measurements can be performed blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Total knee arthroplasty cryo-and compression group (Experimental): use of the cryo- and compression brace during the six postoperative weeks
  Interventions: Device: cryo-and compression brace
- Total knee arthroplasty regular care group (No Intervention): regular care during the six postoperative weeks
- Unicompartmental knee arthroplasty cryo- and compression group (Experimental): use of the cryo- and compression brace during the six postoperative weeks
  Interventions: Device: cryo-and compression brace
- Unicompartmental knee arthroplasty regular care group (No Intervention): regular care during the six postoperative weeks

INTERVENTIONS:
Device: cryo-and compression brace — patients in the intervention groups are instructed to use the cryo- and compression brace during the six postoperative weeks five times a day, for a maximum of 20 minutes. The amount of compression is dependent on a patients' own preference.
  Arms: Total knee arthroplasty cryo-and compression group; Unicompartmental knee arthroplasty cryo- and compression group

SUMMARY:
The goal of this clinical trial is to test the use of a cold and compression brace during the first 6 weeks after surgery in patients who had a total or partial knee replacement.

The main question[s] it aims to answer are:

* What is the effect of the use of cryo- and compression therapy during the first 6 postoperative weeks after knee replacement surgery on pain in rest?
* What is the effect of the use of cryo- and compression therapy during the first 6 postoperative weeks after knee replacement surgery on pain while loading, opioid use, functioning, patient satisfaction and general health, and do participants comply with the therapy?

Participants will be asked to use the cold and compression brace during the six weeks after surgery five times a day, for a maximum of 20 minutes. Researchers will compare with usual care to see the effect on pain, opioid use, functioning, satisfaction and general health.

DETAILED DESCRIPTION:
Total and unicompartmental knee arthroplasty (TKA/UKA) is a widely accepted and effective treatment option for end-stage osteoarthritis (OA) of the knee. Significant long-term improvement in pain, function and quality of life after TKA are reported in literature, yet rehabilitation in the first three months remains challenging. Pain and swelling due to inflammatory reaction after tissue damage may obstruct effective rehabilitation in the early postoperative period. This could result in stiffness of the knee and patient dissatisfaction, also in the long-term. Despite encouraging results after implementing rapid recovery protocols with perioperative local infiltration analgesia and early mobilisation, treatment could still be optimised. Negative side effects (e.g., nausea, vomiting, dizziness) and the increasing abuse of opioid analgesics in modern society drives the search for alternative analgesic techniques. Cryotherapy could play a role in optimising rehabilitation after surgery. Cryotherapy involves the application of cold to the skin surrounding injured soft tissue. Application of cold reduces local blood flow due to vasoconstriction and ensuing the local inflammatory reaction, swelling and heat experience.

The effectiveness of cryotherapy on the recovery after surgery was studied in numerous studies and in the majority - but not in all - of these studies a beneficial effect of the cold therapy was found. Adie et al (2010) show in a systematic review and meta-analysis based on 11 RCT's that using cryotherapy the blood loss is significant lower and the range of motion is higher at discharge. In addition, a small effect on pain is found, cryotherapy leads to lower levels of pain at day 2. This effect was not found at day 1 and 3. No differences were found in complications, analgesics use, length of stay and swelling. Functioning was only measured in one study, so no conclusions could be drawn about that variable. These authors concluded that using cryotherapy postoperatively after a TKA might have benefits, but that the clinical relevance was uncertain. A more recent review performed by Ni et al (2015) confirmed, based on 12 studies, the beneficial results concerning blood loss and pain reduction on day 2. Also, no complications were documented related to the cryotherapy.

Sadoghi et al. (2018) focused on the effects of cryotherapy starting in the first postoperative week and found significant beneficial effects on pain on day 2 and knee flexion on day 6. They did not evidence significant effects in use of analgesics. By contrast, Thijs et al. (2019) found that patients in the cryotherapy group used 2.6 times less opioids as an escape medication during the first four postoperative days compared to the control group. Despite a significant reduction in NRS pain scores before and after cooling in the cryotherapy group, no clear differences on pain between the two groups in the first postoperative week were found. In the long-term too - 2, 6 and 12 weeks postoperatively - no differences could be evidenced. Our recently published RCT has shown that computer-assisted cryotherapy during the first postoperative week following TKA has beneficial in terms of pain reduction and diminished opioid consumption during this first week. At 6 weeks no differences in pain were found. Also the physical examination tests - aROM, knee circumference and Timed Up and Go - showed no difference between groups after 6 weeks. A period of only one week cooling postoperatively can be a reason for short term beneficial effect of the cryotherapy. To our knowledge, no study has been conducted on the effects of 6 weeks cryo and compression therapy after a TKA and UKA.

There are several ways to apply cryotherapy, using ice or cold packs, or mechanical devices which create a standardized cooling treatment of the injured tissue, with and without compression. A review of the currently available literature in TKA and UKA patients stated that standardized continuous cold flow with compression was associated with better outcomes. However, since the financial aspect is also a major element in patient care, cost-effectiveness must be considered as well. Cost benefit analyses demonstrated that simpler devices as ice bag compression bandages or cold packs are far less costly, with no disadvantage in outcomes in several studies. This makes that in the current study an easy-to-use brace with an inserted cold pack, that can be applied with a close fit to the knee, with optional application of manual compression will be used. The combination of cold and compression was suggested to result in longer and improved anaesthetic effect after application.

Primary objective:

Investigating the effect of the use of cryo- and compression therapy during the first 6 postoperative weeks after surgery (TKA en UKA) on pain in rest.

Secondary objective:

Investigating the effect of the use of cryo- and compression therapy during the first 6 postoperative weeks after TKA/UKA surgery on pain while loading, opioid use, functioning, self-perceived change in pain, patient satisfaction and general health. Also the compliance with the cold- and compression therapy will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for a primary TKA or UKA in the Martini Hospital.
* Age ≥ 18 years

Exclusion Criteria:

* per-operative switch from UKA to TKA (only applicable for the UKA patients),
* revision TKA implant (only applicable for the TKA patients),
* rheumatoid arthritis,
* other co-morbidities on which cooling may have a negative effect on (based on judgement of the orthopaedic surgeon),
* inability to read and understand the Dutch language.

Because the cool pack needs to be cooled in a freezer, it is required that a patient or the nursing home has a freezer that can be used.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2023-05-25 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
NRS pain in rest | 6 weeks postoperative
  the NRS pain in rest will be assessed as an important measure of pain

SECONDARY OUTCOMES:
NRS pain in rest | at baseline, daily during first 6 weeks after surgery and at 6 and 12 months
  the NRS pain in rest will be assessed as an important measure of pain
NRS pain during loading | at baseline, daily during first 6 weeks after surgery, 6 weeks postoperative, and at 6 and 12 months
  the NRS pain during loading will be assessed as an additional measure of pain
opioid use | daily during first 6 weeks after surgery
  the amount of opioid use in case of excessive pain
KOOS questionnaire (minus sport and recreation domain) | at baseline and 6 weeks after surgery
  measure of symptoms of the knee
WORQ | at baseline and 6 weeks after surgery
  measure of work ability (functioning)
active Range of Motion | at baseline and 6 weeks after surgery
  measure of knee motion
knee circumference | at baseline and 6 weeks after surgery
  measure of swelling of the knee
Timed Up and Go | at baseline and 6 weeks after surgery
  measure of functional mobility
KOOS-PS | baseline, and 6 and 12 months after surgery
  measure of symptoms of the knee
Oxford Knee score | baseline, and 6 and 12 months after surgery
  measure of symptoms of the knee
EQ-5D 5L | baseline, and 6 and 12 months after surgery
  measure of general health status
Frequency of the use of the cryo and compression brace | daily during first 6 weeks after surgery
  Compliance with cryo- and compression therapy
NRS satisfaction | 6 weeks postoperative, 6 and 12 months after surgery
  patient's satisfaction with the outcome after surgery
achor question: patient perceived change in pain | 6 weeks postoperative, 6 and 12 months after surgery
  the degree in which a patient experiences an improvement in pain compared to baseline (7 point Likert scale)
achor question: patient perceived change in functioning | 6 weeks postoperative, 6 and 12 months after surgery
  the degree in which a patient experiences an improvement in functioning compared to baseline (7 point Likert scale)
NRS patient satisfaction cryo and compression therapy | 6 weeks postoperative
  only for the intervention groups: satisfaction with the use and effectiveness of the intervention

OTHER OUTCOMES:
Complications using the cold compression brace | The first 6 postoperative weeks
  Documentation of complications related to the use of the cold compression brace, including the risk of frostbite and other inconveniences.
Complications using the cold compression brace | Time frame: during the first postoperative year
  Documentation of complications after surgery (infections, re-operations)

CONTACTS AND LOCATIONS:
Overall Officials: Reinoud W. Brouwer, MD PhD, Principal Investigator — Martini Hospital: Martini Ziekenhuis
Locations (1):
- Martini ziekenhuis, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Only deidentified data will be available upon reasonable written request in conjunction with appropriate data use agreement.

REFERENCES:
- [Background] Adie S, Naylor JM, Harris IA. Cryotherapy after total knee arthroplasty a systematic review and meta-analysis of randomized controlled trials. J Arthroplasty. 2010 Aug;25(5):709-15. doi: 10.1016/j.arth.2009.07.010. Epub 2009 Sep 2. PMID 19729279
- [Background] Bourne RB, McCalden RW, MacDonald SJ, Mokete L, Guerin J. Influence of patient factors on TKA outcomes at 5 to 11 years followup. Clin Orthop Relat Res. 2007 Nov;464:27-31. doi: 10.1097/BLO.0b013e318159c5ff. PMID 17891041
- [Background] Holm B, Kristensen MT, Bencke J, Husted H, Kehlet H, Bandholm T. Loss of knee-extension strength is related to knee swelling after total knee arthroplasty. Arch Phys Med Rehabil. 2010 Nov;91(11):1770-6. doi: 10.1016/j.apmr.2010.07.229. PMID 21044725
- [Background] Levy N, Quinlan J, El-Boghdadly K, Fawcett WJ, Agarwal V, Bastable RB, Cox FJ, de Boer HD, Dowdy SC, Hattingh K, Knaggs RD, Mariano ER, Pelosi P, Scott MJ, Lobo DN, Macintyre PE. An international multidisciplinary consensus statement on the prevention of opioid-related harm in adult surgical patients. Anaesthesia. 2021 Apr;76(4):520-536. doi: 10.1111/anae.15262. Epub 2020 Oct 7. PMID 33027841
- [Background] Sadoghi P, Hasenhutl S, Gruber G, Leitner L, Leithner A, Rumpold-Seitlinger G, Kastner N, Poolman RW, Glehr M. Impact of a new cryotherapy device on early rehabilitation after primary total knee arthroplasty (TKA): a prospective randomised controlled trial. Int Orthop. 2018 Jun;42(6):1265-1273. doi: 10.1007/s00264-018-3766-5. Epub 2018 Jan 22. PMID 29356932
- [Background] Thijs E, Schotanus MGM, Bemelmans YFL, Kort NP. Reduced opiate use after total knee arthroplasty using computer-assisted cryotherapy. Knee Surg Sports Traumatol Arthrosc. 2019 Apr;27(4):1204-1212. doi: 10.1007/s00167-018-4962-y. Epub 2018 May 3. PMID 29725749
- [Background] Brouwers HFG, de Vries AJ, van Zuilen M, van Kouswijk HW, Brouwer RW. The role of computer-assisted cryotherapy in the postoperative treatment after total knee arthroplasty: positive effects on pain and opioid consumption. Knee Surg Sports Traumatol Arthrosc. 2022 Aug;30(8):2698-2706. doi: 10.1007/s00167-021-06568-x. Epub 2021 Apr 26. PMID 33903923
- [Background] Ni SH, Jiang WT, Guo L, Jin YH, Jiang TL, Zhao Y, Zhao J. Cryotherapy on postoperative rehabilitation of joint arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2015 Nov;23(11):3354-61. doi: 10.1007/s00167-014-3135-x. Epub 2014 Jun 14. PMID 24928371
- [Background] Chughtai M, Sodhi N, Jawad M, Newman JM, Khlopas A, Bhave A, Mont MA. Cryotherapy Treatment After Unicompartmental and Total Knee Arthroplasty: A Review. J Arthroplasty. 2017 Dec;32(12):3822-3832. doi: 10.1016/j.arth.2017.07.016. Epub 2017 Jul 21. PMID 28802778
- [Background] Schinsky MF, McCune C, Bonomi J. Multifaceted Comparison of Two Cryotherapy Devices Used After Total Knee Arthroplasty: Cryotherapy Device Comparison. Orthop Nurs. 2016 Sep-Oct;35(5):309-16. doi: 10.1097/NOR.0000000000000276. PMID 27648792
- [Background] Thienpont E. Does advanced cryotherapy reduce pain and narcotic consumption after knee arthroplasty? Clin Orthop Relat Res. 2014 Nov;472(11):3417-23. doi: 10.1007/s11999-014-3810-8. Epub 2014 Jul 25. PMID 25059851
- [Background] Soffin EM, YaDeau JT. Enhanced recovery after surgery for primary hip and knee arthroplasty: a review of the evidence. Br J Anaesth. 2016 Dec;117(suppl 3):iii62-iii72. doi: 10.1093/bja/aew362. PMID 27940457
- [Background] Martin SS, Spindler KP, Tarter JW, Detwiler KB. Does cryotherapy affect intraarticular temperature after knee arthroscopy? Clin Orthop Relat Res. 2002 Jul;(400):184-9. doi: 10.1097/00003086-200207000-00023. PMID 12072761
- [Background] Smith J, Stevens J, Taylor M, Tibbey J. A randomized, controlled trial comparing compression bandaging and cold therapy in postoperative total knee replacement surgery. Orthop Nurs. 2002 Mar-Apr;21(2):61-6. doi: 10.1097/00006416-200203000-00009. PMID 11949239
- [Derived] de Vries AJ, Aksakal HK, Brouwer RW. Effects of 6 weeks of cryotherapy plus compression therapy after total or unicompartmental knee arthroplasty: protocol for a single-centre, single-blind randomised controlled trial. BMJ Open. 2024 Jan 29;14(1):e077614. doi: 10.1136/bmjopen-2023-077614. PMID 38286686